CLINICAL TRIAL: NCT01135251
Title: A Double Blind, Parallel-group, Randomized Placebo Controlled, Multicentre Exploratory Study of Dimiracetam in Treatment Induced Painful Neuropathy in Patients With HIV Infection
Brief Title: Safety and Preliminary Evidence of Efficacy of Escalating Doses of Dimiracetam in AIDS Patients With Painful Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotune AG (Industry)
Collaborators: Cross Research S.A. (Industry); Triclinium clinical trial project managment LTD (Unknown)
Responsible Party: Ruggero G Fariello, MD, Chief Medical Officer, Neurotune AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-08-94/NT-11624/003
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: Neuropathy; AIDS
Keywords: Neuropathic pain; AIDS; Dimiracetam; Treatment related painful neuropathy in AIDS patients
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Neuralgia | interventions — dimiracetam; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dimiracetam (Experimental): Capsules containing 400 mg of dimiracetam will be administered orally, twice a day for 8 weeks in ascending schedule, contingent on tolerability of the previous dose, as follows: 1 capsule for two weeks (800mg/day), two capsules for the next two weeks (1600mg/day)and 4 capsules for the final 4 weeks (3200mg/day).
  Interventions: Drug: dimiracetam
- sugar pill (Placebo Comparator): capsules containing 400 mg of inert material will be orally administered twice a day with the same modalities used for the dimiracetam arm: one capsule for 2 weeks, 2 capsules for another 2 weeks and 4 capsules for 4 weeks
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: dimiracetam — 400 mg capsules for oral use to be administered twice a day for a total of 8 weeks
  Arms: dimiracetam
Drug: sugar pill — capsules containing 400 mg of inert material will be orally administered twice a day, one pill for 2 weeks, 2 pills for other 2 weeks and 4 pills for the last 4 weeks.
  Arms: sugar pill

SUMMARY:
One hundred consenting AIDS patients suffering from treatment induced painful neuropathy will be blindly randomize to Active and Placebo groups (ratio A/P = 3/2 and will receive increasing oral doses of dimiracetam starting from 400 mg b.i.d. and doubling the dose every two weeks until a maximum of 1600 mg b.i.d. Escalation to the the higher dose is allowed only if the previous dose did not cause tolerability problems. The highest reached dose will be maintained for a total of 8 week treatment. Patients must have a self evaluated pain of at least 4 on a 10 cm visual analog scale (VAS). Primary end point of the study will be the number of Adverse Events (AEs) reported in the placebo versus the active group. Preliminary evidence of efficacy will be sought by comparing active and placebo group as to the intensity of their pain at study onset and at study end. The pain will be evaluated by the VAS the Total Symptoms Score and the Clinical Global Impression

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 18-65 years;
* females of child-bearing potential only if using a medically accepted method of contraception with a second method of birth control, medically prescribed intrauterine device (IUD), or double barrier method (condom in combination with spermicidal) prior to screening and agreeing to continue its use during the whole duration of the study;
* HIV-positive patients treated with ARTs;
* CD4+ cell count > 200/L at the screening;
* patients affected by neuropathic pain caused by ARTs;
* naïve neuropathic patients or non-responders (residual pain ≥40 mm on the VAS) to standard neuropathy treatments. Drugs for neuropathic pain (NP) must be stopped at screening visit;
* pain intensity ≥40 mm on the VAS at screening;
* pain intensity ≥40 mm on the VAS as the mean of the values collected on the last 4 days prior to the start of treatment (baseline VAS);
* life expectancy of at least 6 months;
* ability to comprehend the full nature and purpose of the study, including possible risks and side effects;
* ability to co-operate with the Investigator or designee and to comply with the requirements of the entire study;
* signed written informed consent prior to inclusion in the study

Exclusion Criteria:

* pregnant or lactating females;
* patients with neuropathic pain due to other factors than the ARTs; any clinically significant underlying disease, according to the Investigator's clinical judgement;
* history of psychosis (e.g. schizophrenia or psychotic depression) or major depression ;
* any current axis I diagnosis including dementia, depression, psychosis, anxiety disorders, mental retardation;
* participation in the evaluation of any investigational drug within 3 months prior to screening (6 months in the neuropathic pain). Use of an investigational drug other than dimiracetam during the study is not permitted;
* treatment with neurostimulating devices such as spinal cord stimulation (SCS), acupuncture, homeopathic remedies for pain or any kind of surgical treatment or blockade for the pain in the 4 weeks prior to screening;
* treatment with any drug for neuropathic pain (NP) after the screening visit; requirement of more than 2 transfusions / month to achieve haemoglobin level > 8 g/dL;
* history of alcohol abuse (defined according to USDA dietary guidelines) or drug abuse during the last 3 months prior to screening;
* history of allergic response to neuropathic treatments or history of anaphylaxis or allergic reactions to drugs in general;
* any abnormality that the Investigator deems to be clinically relevant, either on medical history, physical examination, ECG or in diagnostic laboratory test;
* subjects likely to be non-compliant or uncooperative during the study according to the Investigator or designee's judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
safety and preliminary evidence of efficacy | August 2010

CONTACTS AND LOCATIONS:
Overall Officials: Ruggero G Fariello, MD FAAN, Study Director — Neurotune AG; Daniel R Malan, MD, Principal Investigator — Triple Research, Port Elizabeth SA
Locations (1):
- Aurora Hospital Triple Research, Port Elizabeth, South Africa